CLINICAL TRIAL: NCT06062355
Title: Phase I Clinical Study to Evaluate the Safety, Pharmacokinetics and Radiation Dosimetry of HRS-9815 for PET/CT Imaging in Patients With Prostate Cancer.
Brief Title: Phase I Clinical Study of HRS-9815 for PET/CT Imaging in Patients With Prostate Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-9815-101
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-9815 injection (Experimental)
  Interventions: Drug: HRS-9815 injection

INTERVENTIONS:
Drug: HRS-9815 injection — HRS-9815 injection

SUMMARY:
The study is being conducted to evaluate the the safety, pharmacokinetics, radiation dosimetry of HRS-9815 for PET/CT imaging in adult patients with prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in this clinical trial, understanding of the study procedures and being able to sign the informed consent form in writing;
2. Male, age ≥18 years;
3. ECOG score 0 - 1;
4. Histologically confirmed adenocarcinoma of the prostate;

Exclusion Criteria:

1. Severe urinary incontinence, hydronephrosis, severe micturition dysfunction, etc. Note: Subjects with bladder outflow obstruction or urinary incontinence that can be controlled by the best available standard of care (including pads, drainage, etc.) are eligible to participate in the study.
2. Active syphilis infection.
3. Known allergy, hypersensitivity, or contraindication to the trial product or any component of its formulation.。
4. Active in other clinical studies or less than 4 weeks after the last dose in the previous clinical study at the time of the first dose.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of AEs and SAEs, | up to 30 days follow-up

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | up to 1 days follow-up
time to maximum plasma concentration (Tmax) | up to 1 days follow-up
biological half-life (t1/2) | up to 1 days follow-up
cumulative urinary excretion rate based on radioactivity; | up to 1 days follow-up
Absorbed dose and effective dose of radioactive internal irradiation of the whole body and major organs; | up to 1 days follow-up
Mean standardized uptake value (SUVmean) | up to 1 days follow-up
Maximum standardized uptake value (SUVmax), | up to 1 days follow-up
Tumor-to-background ratio (TBR) [Time Frame: up to 1 days follow-up] | up to 1 days follow-up

IPD SHARING:
Plan to Share IPD: Undecided